CLINICAL TRIAL: NCT05533619
Title: Analysis of Risk Factors of Proton Pump Inhibitor Related Acute Kidney Injury in Hospitalized Patients and Developments of Machine Learning Model
Brief Title: Risk Factors and Machine Learning Model for Proton Pump Inhibitor Related Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xiao Li，MD, Associate professor of pharmacy, Qianfoshan Hospital
Other Study IDs: LCYY-LX-20220104
Record Dates: First submitted 2022-09-02; First posted 2022-09-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Proton Pump Inhibitor; Acute Kidney Injury
Keywords: Proton pump inhibitor; Acute kidney injury; Pharmacoepidemiology; Miss diagnosis; Risk factors; Logic regression
MeSH Terms: conditions — Acute Kidney Injury | interventions — Proton Pump Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI Group
  Interventions: Drug: Proton pump inhibitor
- Non-AKI Group
  Interventions: Drug: Proton pump inhibitor

INTERVENTIONS:
Drug: Proton pump inhibitor — Inpatients using proton pump inhibitor

SUMMARY:
Recent evidence concerns acute kidney injury (AKI) following proton pump inhibitor (PPI) application. Few actual studies have compared the incidence, risk factors, and predictive models of AKI associated with PPI. The present study was a single-center retrospective study. The researchers retrospectively analyzed data from patients who received PPI medications between January 2018 and December 2020. PPI drugs included omeprazole, esomeprazole, rabeprazole, and pantoprazole. The primary outcome of the study was AKI, as defined by kidney disease: improving global outcomes (KDIGO). Secondary outcomes included length of hospital stay, hospital costs, and continuous renal replacement therapy. Independent risk factors associated with AKI were identified by univariate analysis and multifactorial logistic regression analysis (P < 0.05). Logistic regression models were constructed based on the variables obtained from the analysis. Internal validation of the model was performed by the ten-fold cross-validation method. Model discriminatory power was assessed by the area under the curve (AUC) of the receiver operating characteristic curve (ROC). The study aims to develop a PPI-related AKI prediction model based on an electronic medical record system that can be used to predict AKI in hospitalized patients and contribute to the early prevention, diagnosis and treatment of AKI, ultimately reducing morbidity and improving prognosis.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients who used proton pump inhibitor during hospitalization
* Hospital stay ≥ 48h
* Age ≥18 years
* There are two or more blood creatinine tests during hospitalization

Exclusion Criteria:

* Hospital stay < 48h
* Age <18 years
* Glomerular filtration rate (GFR)< 30ml/min/1.73m2 within 48 hours after admission
* AKI was diagnosed on admission
* Less than two Scr test results during hospitalization
* The Scr values were always lower than 40 μmol/L during hospitalization
* Cases with incomplete medical history information

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were included if received treatment with proton pump inhibitor and discharged from the hospital between January 1, 2018 and December 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The incidence of acute kidney injury in hospitalized patients treated with proton pump inhibitors | Through study completion，up to half a year.
  To analyze the incidence of acute kidney injury in hospitalized patients after using proton pump inhibitors, and to build a prediction model. To assess the risk factors before using proton pump inhibitors is helpful to the early prevention, diagnosis and treatment of AKI.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao Li，MD, Jinan, Shandong, China